CLINICAL TRIAL: NCT06235151
Title: Phase 3, Multi-Center, Open-label Study to Test the Diagnostic Performance of Copper Cu 64 PSMA I&T PET/CT in Staging Men With Newly Diagnosed Unfavorable Intermediate-risk, High-risk or Very High-risk Prostate Cancer Electing to Undergo Radical Prostatectomy With Pelvic Lymph Node Dissection
Brief Title: Copper Cu 64 PSMA I&T PET Imaging in Men With Newly Diagnosed Prostate Cancer
Acronym: Solar-Stage
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Curium US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CURCu64PSM0003
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: PSMA; Prostate Cancer; Initial Staging; Solar-Stage; Cu-64 PSMA; PET; Solar
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic Imaging with Copper Cu 64 PSMA I&T (Experimental): Copper Cu 64 PSMA I&T Injection
  Interventions: Drug: Copper Cu 64 PSMA I&T

INTERVENTIONS:
Drug: Copper Cu 64 PSMA I&T — Radiopharmaceutical PET imaging tracer injected intravenously for staging of prostate cancer.

SUMMARY:
This is a prospective, open-label Phase 3 study to evaluate copper Cu 64 PSMA I&T injection for PET/CT imaging in patients with newly diagnosed unfavorable intermediate high-risk, high-risk or very high-risk prostate cancer.

DETAILED DESCRIPTION:
The study will include approximately 323 patients with newly diagnosed unfavorable intermediate high-risk, high-risk or veru high-risk prostate cancer electing to undergo radical prostatectomy with pelvic lymph node dissection. Each patient will be administered an 8 mCi (± 10 percent) intravenous dose of copper Cu 64 PSMA I&T injection. PET/CT imaging will be acquired for all patients at 1-4 hours ± 15 minutes post copper Cu 64 PSMA I&T injection.

The PET/CT images will be interpreted independently by three readers blinded to all patient information. Each patient study will be assessed and scored for the detection of lesions considered positive for Prostate Cancer (PC) in pelvic lymph nodes. Positive lesions in the prostate, extra pelvic lymph nodes, bones and soft tissue/viscera will also be recorded. Analysis of the reads will be used for determination of sensitivity and specificity of copper Cu 64 PSMA I&T PET/CT by comparison to the reference standard of histopathology after matching by hemipelvis with at least one true positive lesion defining a true positive patient. Detection of PC outside the pelvis on the copper Cu 64 PSMA I&T PET/CT will be assessed using reference standard of histopathology and if not available conventional imaging. Baseline conventional imaging will be reviewed for PC disease or no disease by independent radiology readers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven prostate adenocarcinoma.
* Planned prostatectomy with pelvic lymph node dissection.
* Unfavorable intermediate-risk, high-risk, or very high-risk disease defined by NCCN Guidelines Version 1.2023 and previous versions.
* Male aged greater than or equal to 18 years.
* Able to understand and provide signed written informed consent.

Exclusion Criteria:

* Androgen deprivation therapy, neoadjuvant chemotherapy, radiation therapy (including local ablation techniques), or any investigational therapy against Prostate Cancer (PC) prior to prostatectomy.
* Patients participating in an interventional clinical trial within 30 days and having received an Investigational Product (IP) within five (5) biological half-lives prior to administration.
* Patients with any medical condition or circumstance (including receiving an IP or not capable of having a PET study) that the investigator believes may compromise the data collected or lead to a failure to fulfill the study requirements.
* Patients who are planned to have an x-ray contrast within 24 hours or other PET radiotracer within 10 physical half-lives prior to the PET scan. If Barium contrast is administered this should be cleared before the PET scan.
* Patients who are administered any high energy (greater than 300 KeV) gamma emitting radioisotopes within five (5) physical half-lives prior to copper Cu 64 PSMA I&T administration.
* Patients with known hypersensitivity to the active substance or any of the excipients of the IP.
* Patients who had a PSMA PET scan as part of their standard medical care within 90 days prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 323 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 4 Hours
  Determine the presence of metastatic pelvic lymph nodes relative to histopathology reference standard. At least one positive pelvic lymph node on the PET scan and one positive lymph node as determined by histopathology on the same side of the pelvis (left or right) will be counted a true positive at the patient level.
Specificity | 4 Hours
  Determine the absence of metastatic pelvic lymph nodes relative to histopathology reference standard. Negative pelvic lymph node on the PET scan and negative pelvic lymph nodes as determined by histopathology on the same side of the pelvis (Left or Right) will be counted a true negative at the patient level.

SECONDARY OUTCOMES:
Inter-reader and intra-reader agreement of copper Cu 64 PSMA I&T PET/CT interpretation on a per-patient basis | 4 Hours
  Reader kappa statistics of copper Cu 64 PSMA I&T PET/CT scan interpretation by the blinded independent readers.
Incidence of adverse events in copper Cu 64 PSMA I&T injection | At time of dose administration up to 72 Hours
  Treatment-emergent adverse events (AEs) will be assessed and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

OTHER OUTCOMES:
Determine the relationship of Prostate Specific Antigen (PSA) level, Gleason score, and the diagnostic performance of copper Cu 64 PSMA I&T PET/CT | 4 Hours
  Correlation of sensitivity, specificity, detection rate, and Positive Predictive Value (PPV) to baseline PSA and unfavorable intermediate-risk, high-risk or very high-risk at the time of prostatectomy.
Assess PPV of lesions on copper Cu 64 PSMA I&T PET/CT outside the prostate and pelvic lymph nodes (M1 disease) | 4 Hours
  Proportion of patients with M1 lesions on copper Cu 64 PSMA I&T PET/CT subsequently confirmed to be TP by biopsy, surgery and confirmatory imaging.
Assess the impact of copper Cu 64 PSMA I&T PET/CT on the intended clinical management of study participants | 4 Hours
  Percentage of patients in whom the copper Cu 64 PSMA I&T PET/CT changed the intended patient management (major and other changes).
Assess the detection rate on patient level and split by pelvic lymph nodes and extra pelvic lesions | 4 Hours
  Patient level positivity rates of copper Cu 64 PSMA I&T split by pelvic lymph nodes and extra pelvic lesions.
Determine sensitivity and specificity by risk group (unfavorable intermediate, high, or very high risk) | 4 Hours
  Determine the diagnostic performance of copper Cu 64 PSMA I&T PET/CT for the detection of presence or absence of pelvic lymph node metastasis in pre-prostatectomy patients by risk group (unfavorable intermediate, high, or very high risk).

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Arkansas Urology, Little Rock, Arkansas
  - Providence Medical Foundation, Fullerton, California
  - Tower Urology, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California, Irvine, Orange, California
  - San Francisco VA Medical Center, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Stanford Hospital & Clinics, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami Hospital and Clinics - Sylvester Comprehensive Cancer Center, Miami, Florida
  - CIRA Health, Miami, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Florida Urology Partners, Tampa, Florida
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - Urology of Indiana, LLC, Carmel, Indiana
  - IU Health Neuroscience Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Hospital, Kansas City, Kansas
  - United Theranostics, Glen Burnie, Maryland
  - VA Boston Healthcare System, Boston, Massachusetts
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - John Cochran VA Medical Center, St Louis, Missouri
  - Great Plains Health, Diagnostic Imaging, North Platte, Nebraska
  - XCancer, Omaha, Nebraska
  - United Theranostics, Princeton, New Jersey
  - Adaptive Research Inc., Hawthorne, New York
  - Queens Hospital Center, Jamaica, New York
  - Columbia University Medical Center, New York, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - UNC Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Dayton Physicians Network / Greater Dayton Cancer Center, Kettering, Ohio
  - VA Portland Health Care System, Portland, Oregon
  - Hollings Cancer Center, Charleston, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - The Urology Place, San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No